CLINICAL TRIAL: NCT02277756
Title: Pain Neuromodulation in Adults With Autism Spectrum Disorder
Brief Title: Pain in Adults With Autism Spectrum Disorder
Acronym: DOUPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: autistic recruitment problems
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DOUPA (RB 14.035)
Record Dates: First submitted 2014-10-21; First posted 2014-10-29 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Autism; Pain
Keywords: high functioning autism; endogenous modulation systems
MeSH Terms: conditions — Autistic Disorder; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high functioning Autism (Experimental): Thermal stimulation with test thermode Thermic stimulations (tonic heat pain stimulation and cold-pressor test) are used to test excitatory and inhibitory pain mechanisms with high functioning Autism
  Interventions: Device: thermode
- witness (Placebo Comparator): Thermic stimulations (tonic heat pain stimulation and cold-pressor test) are used to test excitatory and inhibitory pain mechanisms with a witness
  Interventions: Device: thermode

INTERVENTIONS:
Device: thermode — thermal stimulation with test thermode

SUMMARY:
Pain insensibility is often described in people with autism. The aim of this study is to test the pain perception in adults with autistic spectrum disorder without intellectual disability. An experimental model of pain is used to measure endogenous modulation systems. Thermic stimulations (tonic heat pain stimulation and cold-pressor test) are used to test excitatory and inhibitory pain mechanisms. Salivary cortisol and automatic nervous system (heart rate and blood pressure with an electrocardiogram (Brest :system dantec keypoint natus G3 ; Paris: nexfin HD®) are also tested and behavioral response to thermal stimulation assessed by an inspired behavior scale.

DETAILED DESCRIPTION:
Adults with autism without intellectual disability (IQ > 85) are matched with members of siblings and control group (sex and chronological age).

Pain reactivity (Visual analog scale,endogenous modulation systems, salivary cortisol, automatic nervous system and behavioral responses to thermal stimulation assessed by an inspired behavior scale.) in adult with autism is tested using an experimental model of pain. Excitatory and inhibitory modulation systems were elicited using a temporal summation test administered before and after activation of the Diffuse Noxious Inhibitory Control (DNIC) by means of a cold-pressor test.

Demographic and clinical data are also collected (sensory profile, sleep disorders and depression inventory).

ELIGIBILITY:
Non-specific inclusion criteria:

* intellectual quotient >85
* consent form signed

Inclusion Criteria autism group :

* autism diagnosis (CIM 10) from multidisciplinary evaluation (ADI-r, ADOS)
* sibling without autism or developmental disorder

Non-specific Exclusion Criteria:

* chronic pain
* pregnancy, breast feeding
* consent form no signed

Exclusion criteria sibling and witness groups:

- diagnosis of autism or developmental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by Computerized Visual analog scale | one day

SECONDARY OUTCOMES:
salivary cortisol | one day
Behavioral response to thermal stimulation assessed by an inspired EDM-DI behavior scale | one day
heart rate variability | one day

CONTACTS AND LOCATIONS:
Overall Officials: Gildas L'HEVEDER, Doctor, Principal Investigator — CHRU Brest
Locations (1):
- CHRU Brest, Brest, France